CLINICAL TRIAL: NCT00746551
Title: Low Dose Intravenous Versus Oral Iron for Iron Deficiency Anemia Starting Late in Pregnancy: A Randomized Controlled Trial
Brief Title: Intravenous Versus Oral Iron in Late Pregnancy: Results of Treatment
Acronym: EIVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Principal Investigator, Pharuhas Chanprapaph, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 296/2551(EC3)
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Anemia; Pregnancy Complications
Keywords: iron deficiency anemia; pregnancy; third trimester; intravenous iron; efficacy; a randomized trial; Female; Ferric Compounds/therapeutic use*; Infusions, Intravenous; Hematologic/therapy*
MeSH Terms: conditions — Anemia; Pregnancy Complications; Anemia, Iron-Deficiency | interventions — Long-Term Synaptic Depression; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferrous fumarate, Ferri-6®, Oral tablet (Active Comparator): In the O-group, women had to take 3 ferrous fumarate tablets (Ferli-6®) everyday with a total of 200 mg of elemental iron per day from 33 weeks gestation until delivery. Emphasizing and monitoring for compliance to the treatment protocol were carried out.
  Interventions: Drug: Ferli-6® (Continental Pharm co., ltd.)
- iron sucrose, Venofer®, intravenous drug (Experimental): Women in the IV-group received 500 mg iron sucrose (Venofer®, Vifor International AG, St. Gallen, Switzerland) divided into three weekly administrations. Two doses of 200 mg iron sucrose were given at 33 and 34 weeks gestation while the remaining (100 mg) was infused at gestation of 35 weeks. Thereafter, women in this group received no further iron therapy until delivery. In preparation, 200 mg of iron sucrose was diluted into 100 ml of 0.9% saline solution.
  Interventions: Drug: Venofer® (Vifor AG, St. Gallen, Switzerland)

INTERVENTIONS:
Drug: Ferli-6® (Continental Pharm co., ltd.) — In the O-group, women had to take 3 ferrous fumarate tablets (Ferli-6®) everyday with a total of 200 mg of elemental iron per day from 33 weeks gestation until delivery. Emphasizing and monitoring for compliance to the treatment protocol were carried out.
  Arms: Ferrous fumarate, Ferri-6®, Oral tablet
Drug: Venofer® (Vifor AG, St. Gallen, Switzerland) — Women in the IV-group received 500 mg iron sucrose (Venofer®, Vifor International AG, St. Gallen, Switzerland) divided into three weekly administrations. Two doses of 200 mg iron sucrose were given at 33 and 34 weeks gestation while the remaining (100 mg) was infused at gestation of 35 weeks. Thereafter, women in this group received no further iron therapy until delivery. In preparation, 200 mg of iron sucrose was diluted into 100 ml of 0.9% saline solution.
  Arms: iron sucrose, Venofer®, intravenous drug

SUMMARY:
The purpose of this study is to compare the efficacy of body iron storage replenishment between low dose intravenous iron and oral iron in late pregnancy.

DETAILED DESCRIPTION:
Despite routine antenatal oral iron supplementation, the prevalence of iron deficiency anemia (IDA) in the 3rd trimester of pregnancy in developing countries remains high. Apparently, intravenous iron sucrose appears to be safe and efficient in treating within a short period. From literature review, no study of intravenous iron for IDA treatment has been carried out in the third trimester of pregnancy. This research aims to compare the efficacy of body iron storage replenishment at 3 weeks as labor may take place at this point in some women. In this study,500 mg intravenous iron has been given weekly instead of every other day for the sake of patient's convenience in the hope that parenteral iron may become another alternative for treatment of pregnant women with iron deficiency anemia who have difficulties or failures with oral iron.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years old
2. Singleton pregnancy at 32 weeks gestation
3. Having anemia in the third trimester according to World Health Organization, namely, with a hemoglobin level of < 11 g/dL or hematocrit of < 33%
4. Having no underlying disease such as hypertension, gestational diabetes mellitus, heart disease, peptic ulcer, etc.
5. Having no history of allergy to iron containing medication
6. Having no history or other allergic conditions or asthma
7. Having no thalassemia disease, for examples: B thalassemia major, hemoglobin E/ B thalassemia, homozygous hemoglobin E, Hemoglobin H, AE Bart disease, and EF Bart disease. Pregnant women who have iron deficiency anemia and are thalassemia carriers such as A-thalassemia 1, B-thalassemia, or less severe Hb E/ B thalassemia are able to enter the study.
8. Having no history of bleeding tendency
9. Having no history of blood transfusion within the prior 120 days
10. Having no history of delivery before 36 weeks gestation
11. Giving consent and having signed the consent form for this study

Exclusion Criteria:

1. Stool exam revealed parasitic infestation
2. C-reactive protein > 3 mg/L
3. Serum ferritin > 15 mcg/L

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pornpimol Ruangvutilert, MD, PhD., Principal Investigator — Obstetrics and Gynecology Department, Faculty of Medicine Siriraj Hosptial, Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at Maternal Fetal Medicine Unit, Siriraj Hospital between September 2008 and December 2009. Singleton pregnant women aged 18-45 years old at GA of 32 weeks with Hb level < 11.0 g/dL, serum ferritin levels < 15 µg/L and CRP of < 20 mg/L with negative stool examination for parasitic infection were recruited into the study.
Period: At Gestational Age of 36 Weeks
Arm/Group | Iron Sucrose, Venofer®, Intravenous Drug | Ferrous Fumarate, Ferri-6®, Oral Tablet
Started | 40 | 40
Completed | 38 | 36
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4
Period: At Delivery (GA of 39 Weeks)
Arm/Group | Iron Sucrose, Venofer®, Intravenous Drug | Ferrous Fumarate, Ferri-6®, Oral Tablet
Started | 40 | 40
Completed | 25 | 25
Not Completed | 15 | 15
Not completed — Lost to Follow-up | 9 | 7
Not completed — preterm delivery, delivery elesewhere | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Iron Sucrose, Venofer, Intravenous Drug; Ferrous Fumarate, Ferri-6, Oral Tablet: Initially, there were 194 subjects enrolled but 114 cases were excluded from the study. Among those, 104 cases did not meet the inclusion criteria and 10 cases refused to take part. A total of 80 eligible patients were equally randomised and allocated in to 2 groups of intravenous sucrose complex-group (ISC) and oral ferrous fuamrate-group (OFF) . At GA of 36 weeks, there were 4 cases of the OFF-group and 2 cases of the ISC-group lost to follow-up. At delivery, there were 50 patients remained in the study whereas 30 patients were excluded from statistical analysis due to losing to follow-up (16 cases), delivery at other hospitals (10 cases) and preterm deliveries (4 cases).
- Total: Total of all reporting groups
Arm/Group | Iron Sucrose, Venofer, Intravenous Drug | Ferrous Fumarate, Ferri-6, Oral Tablet | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.9) | 24.9 (5.9) | 24.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Body weight [Mean (Standard Deviation); unit: kg] | 48.1 (8.1) | 50.2 (6.6) | 49.2 (7.4)
Body mass index [Mean (Standard Deviation); unit: kg/sq.m] | 19.7 (3.4) | 20.1 (2.2) | 19.9 (2.9)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] | 3.7 (2.0) | 4.0 (2.3) | 3.9 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Serum Ferritin Level
Time Frame: 3 weeks after intervention
Measure: Mean (Standard Deviation); unit: µg/dL
Groups:
- Iron Sucrose, Venofer, Intravenous Drug: Patients in the study group (ISC-group) were given 500 mg of ISC (Venofer®, Vifor International AG, St. Gallen, Switzerland) in three divided doses. The administration was given weekly with the maximum dose of 200 mg from GA 33 to 35 weeks. Thereafter, no other iron supplementation was given to this group until delivery. In preparation, 200 mg of ISC was diluted into 100 ml of 0.9% saline solution. Test dose was performed by slow infusion of 5 ml solution within 5 minutes. This was only required on the first ISC treatment.
  If no adverse reactions were observed in 15 minutes, the remaining solution was infused to the patient within 30 minutes. Subsequent infusions were administered in 40 minutes. Careful post infusion observation was conducted in every case for at least 30 minutes to ensure patient safety.
  Patients in the ISC-group who failed to complete the 3-week treatment course were withdrawn from the trial.
- Ferrous Fumarate, Ferri-6, Oral Tablet: The patients in the control group (OFF-group) were instructed to have 3 oral ferrous fumarate tablets (Ferli-6®, Continental-Pharm, Thailand) daily with a total of 200 mg elemental iron per day until delivery. The remaining of OFF tablets was counted at every visit to evaluate patient compliance. Patients in the OFF-group who took less than 80% of the allocated medication were withdrawn from the trial.
Arm/Group | Iron Sucrose, Venofer, Intravenous Drug | Ferrous Fumarate, Ferri-6, Oral Tablet
Number analyzed (Participants) | 38 | 36
µg/dL | 136.1 (55.0) | 28.3 (14.8)

2. Secondary Outcome: Haemoglobin Level
Time Frame: 3 weeks after intervention
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Iron Sucrose, Venofer, Intravenous Drug | Ferrous Fumarate, Ferri-6, Oral Tablet
Number analyzed (Participants) | 38 | 36
g/dL | 10.6 (0.6) | 10.2 (1.0)

ADVERSE EVENTS:
Groups:
- Iron Sucrose, Venofer®, Intravenous Drug: In preparation, 200 mg of ISC was diluted into 100 ml of 0.9% saline solution. Test dose was performed by slow infusion of 5 ml solution within 5 minutes. This was only required on the first ISC treatment.
  If no adverse reactions were observed in 15 minutes, the remaining solution was infused to the patient within 30 minutes. Subsequent infusions were administered in 40 minutes. Careful post infusion observation was conducted in every case for at least 30 minutes to ensure patient safety.
  Patients in the ISC-group who failed to complete the 3-week treatment course were withdrawn from the trial.
- Ferrous Fumarate, Ferri-6®, Oral Tablet: Patients in the OFF-group who took less than 80% of the allocated medication were withdrawn from the trial.
Arm/Group | Iron Sucrose, Venofer®, Intravenous Drug | Ferrous Fumarate, Ferri-6®, Oral Tablet
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No